CLINICAL TRIAL: NCT06139289
Title: A Review of External Ventricular Drain Placement at the Bedside Versus Operating Room
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 102.MBSI.2022.D
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: External Ventricular Drain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: EVD placements in the OR versus the bedside. — Reducing EVD-related complications
  Other Names: EVD placement environment

SUMMARY:
External ventricular drain (EVD) placement is a common neurosurgical procedure and provides a way to monitor intracranial pressure. EVDs are utilized in the management of a wide array of neurosurgical indications, such as subarachnoid hemorrhage, trauma, intraventricular hemorrhage, cerebrospinal fluid (CSF) leaks, and hydrocephalus.

DETAILED DESCRIPTION:
External ventricular drain (EVD) placement is a common neurosurgical procedure and provides a way to monitor intracranial pressure. EVDs are utilized in the management of a wide array of neurosurgical indications, such as subarachnoid hemorrhage, trauma, intraventricular hemorrhage, cerebrospinal fluid (CSF) leaks, and hydrocephalus. While generally regarded as safe, EVDs are associated with a significant risk of complications, such as hemorrhage, infection, and improper placement resulting in a need for replacement and the patient undergoing an additional procedure.

Significant research has been conducted reducing these complications, with a major focus on issues with the procedure itself, instruments utilized for EVD placement, or post-procedure care of the EVD. To the knowledge, few investigations have focused on the EVD placement environment ( the operating room versus the bedside). Aim to evaluate the circumstances and complications rates associated with EVD placement between these two settings at Methodist Dallas Medical Center (MDMC).

ELIGIBILITY:
Inclusion Criteria:

* • Patients ≥18 years old

  * Any patient undergoing EVD placement at MDMC between January 2018 and August 2022

Exclusion Criteria:

* • Any patient not meeting criteria in section 3.1

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients ≥18 years old Any patient undergoing EVD placement at MDMC between January 2018 and August 2022
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2025-07-21 (Actual)

PRIMARY OUTCOMES:
EVD Placement Success | 30 Days
  development of best-practice recommendations for future EVD placements

CONTACTS AND LOCATIONS:
Overall Officials: Richard Meyrat, MD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Study data or any protected health information will not be shared with anyone that is not delegated to the study. The PI is committed to disseminate research results in a timely fashion. Sharing of results generated by the data analysis during the course of the project will be through presentation at national scientific meetings and/or publication in open access journals. All information obtained will be source de-identified and presented on a large scale and not traceable to any one particular individual.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 2 years

REFERENCES:
- [Background] Foreman PM, Hendrix P, Griessenauer CJ, Schmalz PG, Harrigan MR. External ventricular drain placement in the intensive care unit versus operating room: evaluation of complications and accuracy. Clin Neurol Neurosurg. 2015 Jan;128:94-100. doi: 10.1016/j.clineuro.2014.09.026. Epub 2014 Oct 5. PMID 25436470